CLINICAL TRIAL: NCT00611039
Title: Clinical Pilot, Open, Comparative and Randomized Trial to Evaluate the Efficacy and Security of Darunavir/Ritonavir 900/100 mg Once a Day as an Antiretroviral Treatment Simplification Strategy
Brief Title: Evaluate the Efficacy and Security of Darunavir/Ritonavir 900/100 mg Once a Day as an Antiretroviral Treatment Simplification Strategy
Acronym: DRV900100QD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRV 900100 QD
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: HIV Infections
Keywords: Darunavir/ritonavir; virtual inhibitory quotient; dose reduction
MeSH Terms: conditions — HIV Infections | interventions — Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Darunavir 900mg + ritonavir 100 mg once a day
  Interventions: Drug: Darunavir 900mg + ritonavir 100 mg once a day
- 2 (Active Comparator): Darunavir 600mg + ritonavir 100mg twice day
  Interventions: Drug: Darunavir 600mg + ritonavir 100mg twice day

INTERVENTIONS:
Drug: Darunavir 900mg + ritonavir 100 mg once a day — Darunavir 900mg + ritonavir 100 mg once a day
  Arms: 1
Drug: Darunavir 600mg + ritonavir 100mg twice day — Darunavir 600mg + ritonavir 100mg twice day
  Arms: 2

SUMMARY:
Basing in studies which have related the darunavir (DRV) virtual inhibitory quotient (vIQ) with the virological response, it is possible to think in the possibility of simplifying the rescue treatment with DRV/ritonavir to 900/100 mg once a day in those patients who are being treated with DRV/ritonavir 600/100 mg twice a day and who, besides having undetectable viral load, have a vIQ over 2. This strategy would not jeopardize the efficacy of the antiretroviral treatment and would have less impact in the lipid profile of the patients as well as less pharmaceutical expenditure.

DETAILED DESCRIPTION:
The probability of achieving viral replication suppression during the treatment with DRV has been related to both the extent of viral resistance to DRV (inhibitory concentration 50%, IC50) and the drug concentration. Moreover, the DRV virtual inhibitory quotient (vIQ) has been related significantly with the virological response to DRV treatment. So patients with a DRV vIQ >= 1,5 had a 8-times higher probability of having viral load < 50 copies/mL after 24 weeks of treatment than those having a vIQ < 1,5.

Considering the previous arguments, it is possible to think in the possibility of simplifying the rescue treatment with DRV/ritonavir to 900/100 mg once a day in those patients who are being treated with DRV/ritonavir 600/100 mg twice a day and who, besides having undetectable viral load, have a DRV vIQ over 2. This strategy would not jeopardize the efficacy of the antiretroviral treatment and would have less impact in the lipid profile of the patients as well as less pharmaceutical expenditure.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years.
2. HIV-infected patients.
3. Stable antiretroviral treatment including darunavir/ritonavir 600/100 every 12 hours for at least 4 weeks.
4. HIV viral load < 50 copies/mL for at least 12 weeks.
5. Resistance test (Genotype or Virtual Phenotype) before starting tipranavir treatment.
6. Darunavir vIQ >= 2.
7. Subject able to follow the treatment period.
8. In women, negative pregnancy test or not in fertile age (defined as at least one year from menopause or undergoing any surgical sterilisation technique), or undertaking to use a barrier contraceptive method during the study.
9. Signature of the informed consent.

Exclusion Criteria:

1. AIDS-defining illness in the last 4 weeks.
2. Suspicion of unsuitable antiretroviral treatment compliance.
3. In women, pregnancy or breastfeeding.
4. Record or suspicion of incapability to cooperate as appropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HIV-1 viral load < 50 copies /mL | Basal, week 2, week 4, week 8, week 12 ,week 24week 36 and week 48

SECONDARY OUTCOMES:
DRV plasma trough concentration | Screening, Basal, week 2, week 4, week 8, week 12, week 24, week 36 and week 48
DRV Virtual inhibitory quotient (vIQ) | Screening, Basal, week 2, week 4, week 8, week 12, week 24, week 36 and week 48
CD4 and CD8 lymphocytes count | Screening, Basal, week 12, week 24, week 36 and week 48
Physical examination including weight and height | Screening, Basal, week 2, week 4, week 8, week 12, week 24, week 36 and week 48
Karnofsky index | Screening, Basal, week 2, week 4, week 8, week 12, week 24, week, 36 and week 48
Adverse events | Screening, Basal, week 2, week 4, week 8, week 12, week 24, week 36 and week 48
Lipid profile (total cholesterol, HDL-cholesterol. LDL-cholesterol and triglycerides) | Screening, Basal, week 2, week 4, week 8, week 12, week 24, week 36 and week 48
Treatment adherence (assessed by the physician, but not recovered in the data base) | Screening, Basal, week 2, week 4, week 8, week 12, week 24, week 36 and week 48
Genotype, if virological failure occurs | When virological failure

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Clotet, MD,PhD, Principal Investigator — Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain

REFERENCES:
- [Derived] Molto J, Valle M, Santos JR, Mothe B, Miranda C, Cedeno S, Negredo E, Yritia M, Videla S, Barbanoj MJ, Clotet B. Treatment simplification to once daily darunavir/ritonavir guided by the darunavir inhibitory quotient in heavily pretreated HIV-infected patients. Antivir Ther. 2010;15(2):219-25. doi: 10.3851/IMP1519. PMID 20386077